CLINICAL TRIAL: NCT03686683
Title: A Randomized Phase 3, Open-Label Trial of Sipuleucel-T Administered To Patients On Active Surveillance For Newly Diagnosed Prostate Cancer
Brief Title: Open- Label Trial of Sipuleucel-T Administered to Active Surveillance Patients for Newly Diagnosed Prostate Cancer
Acronym: ProVent
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dendreon (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P17-1; ProVent (Other: Dendreon Pharmaceuticals LLC)
Record Dates: First submitted 2018-09-25; First posted 2018-09-27 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2023-10

CONDITIONS: Adenocarcinoma of the Prostate
Keywords: ISUP Grade Group 1 or 2; Number biopsies 1 or >1 (≤12 months of Screening)
MeSH Terms: interventions — sipuleucel-T

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 2:1 to the sipuleucel-T arm or the control arm.Participants randomized to sipuleucel-T arm will receive 3 infusions of sipuleucel-T at approximately 2-week intervals. Participants randomized to the control arm will be followed on AS as standard of care described in the schedule of events.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group: Sipuleucel-T (Experimental): Sipuleucel-T is an autologous cellular immunotherapy available as a suspension for intravenous infusion. Participants randomized to sipuleucel-T arm will receive 3 infusions of sipuleucel-T at approximately 2-week intervals.
  Interventions: Biological: sipuleucel-T
- Control Arm: Active Surveillance (No Intervention): Participants randomized to the control arm will be followed on Active Surveillance described in the schedule of events.

INTERVENTIONS:
Biological: sipuleucel-T — Sipuleucel-T is an autologous cell product consisting of antigen presenting cells (APCs) loaded with recombinant fusion protein composed PAP linked to GM-CSF (PA2024), a recombinant fusion protein composed of prostatic acid phosphatase (PAP), linked to granulocyte-macrophage colony-stimulating factor (GM-CSF).
  Arms: Treatment Group: Sipuleucel-T

SUMMARY:
The ProVent study is a randomized, open-label study designed to assess the efficacy of sipuleucel-T in reducing the progression of lower risk non-metastatic prostate cancer compared to participants followed on active surveillance as standard of care.

DETAILED DESCRIPTION:
The ProVent Study is designed to look at participants who receive sipuleucel-T compared to control participants followed on active surveillance (AS). The study will enroll participants being followed by AS and initially diagnosed within 12 months prior to Screening with either International Society of Urological Pathology (ISUP) Grade Group 1 or 2 adenocarcinoma of the prostate.

The Screening Phase will begin at the completion of the informed consent process and continues until randomization. After Screening assessments are completed, eligible participants will be randomized 2:1 to the sipuleucel-T arm or the control arm. Participants randomized to sipuleucel-T arm will receive product as described in the sipuleucel-T approved label.

Participants will undergo their first leukapheresis within 60 days of randomization.

Participants randomized to the control arm will be followed on AS. The Active Phase will begin at randomization and continues through completion of the end of Active Phase study visit (within 30 days of Biopsy 2). Once a Participant from either the sipuleucel-T or control arms completes the end of Active Phase visit, they will enter the Follow-up Phase and complete Follow-up Phase visits every 6 months starting from their last Active Phase visit. The Follow-up Phase visits end when the last Participant enrolled completes Biopsy 2 and end of Active Phase visit or until the study is terminated by the sponsor.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age is ≥ 18 years
* 2. Written informed consent provided prior to the initiation of study procedures
* 3. Histologically proven adenocarcinoma of the prostate initially diagnosed ≤12 months of Screening. All biopsy slides with participant information redacted must be submitted for blinded independent central review (BICR).
* 4. Prostate cancer diagnosis determined by BICR as one of the following: 4a. ISUP Grade Group 1 with 3 or more cores positive from a systematic (≥10 cores) biopsy 4b. ISUP Grade Group 1 with ≥ 1 core positive with ≥50% cancer involvement from a systematic (≥10 cores) biopsy 4c. ISUP Grade Group 1 from 3 or more positive cores from any combination of cores from a systematic (≥10 cores) biopsy and MRI targeted biopsy (note: multiple cores from each MRI targeted lesion will count as 1 core) 4d. ISUP Grade Group 1 from a negative systematic (≥10 cores) biopsy and an MRI targeted core positive with ≥50% cancer involvement 4e. ISUP Grade Group 2 from a systematic (≥10 cores) biopsy with <50% of the total number of any cores positive for cancer 4f. ISUP Grade Group 2 from a negative systematic (≥10 cores) biopsy and MRI targeted core(s) positive for Gleason 3+4 (see note below) 4g. ISUP Grade Group 2 from any combination of cores from a systematic (≥10 cores) biopsy and MRI targeted biopsy (see note below)

Note for 4f and 4g: the total number of positive cores must be <50% of total cores from both the systematic biopsy and MRI targeted lesions; each MRI targeted lesion, irrespective of multiple positive cores, will each count as 1 core for the total number of positive cores, e.g., 4 targeted lesions with 2 positive cores each will only add 4 to the total core count.

* 5. Participant consents to standard of care for biopsy frequency of 2 on-study prostate biopsies and to provide biopsy tissue for study endpoint analysis.
* 6. Estimated life expectancy ≥ 10 years
* 7. Candidate for primary curative therapy (e.g., surgery or radiation) if prostate cancer progression occurs
* 8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* 9. Adequate baseline hematologic, renal, and liver function tests as evidenced by laboratory test results within the following ranges ≤30 days prior to randomization White blood cell (WBC) count ≥ 3.0 x 10^6 cells/mL Absolute neutrophil count (ANC) ≥ 1.5 x 10^6 cells/mL Platelet count ≥ 1.0 x10^5 cells/uL Hemoglobin (Hgb) ≥ 10.0 g/dL Creatinine ≤ 1.5 mg/dL Total bilirubin ≤ 1.5 x upper limit of normal (ULN) Alanine aminotransferase (ALT) ≤ 2.0 x ULN Aspartate aminotransferase (AST) ≤ 2.0 x ULN

Exclusion Criteria:

* 1. Former therapy for prostate cancer (local or systemic)
* 2. Any previous prostatic surgical procedure that significantly changes the anatomy of prostate (at the discretion of sponsor's Medical Monitor)
* 3. Any investigational product received for prostate cancer
* 4. Prostate biopsy specimen reveals neuroendocrine or small cell features
* 5. Primary Gleason score is ≥ 4 or any Gleason pattern 5
* 6. Any evidence of locally advanced, regional or metastatic disease, including regional and distant lymph node enlargement (Nodes ≥1.5 cm in the short axis are considered pathologic and measurable)
* 7. A history of a cerebrovascular event (CVE) or transient ischemic attack (TIA)
* 8. Participant has used a 5-alpha-reductase inhibitor (e.g., finasteride or dutasteride) continuously for ≥ 6 months and within 6 months prior to study Screening
* 9. Participant has a history of any other stage I-IV malignancy, except for basal or squamous cell skin cancer. The Participant must be disease free and off any malignancy-related treatment for at least 5 years.
* 10. Participant has prior use within 30 days of study Screening of any herbal, dietary, or alternative anti-cancer treatment or product, such as PC-SPES (or PC-x product), saw palmetto, ketoconazole, an estrogen-containing nutraceutical, or high dose calcitriol (>0.5 μg/day). The Investigator will consider herbal therapies on a case-by-case basis to determine whether they fall into the category of prohibited medications based on their potential for hormonal or anti-cancer or anti-cancer properties.
* 11. Need for systemic chronic immunosuppressive therapy (e.g., anti-tumor necrosis factor alpha monoclonal antibodies, glucocorticoids)
* 12. Uncontrolled, concurrent illness including, but not limited to the following: ongoing or active infection (bacterial, viral, or fungal), symptomatic congestive heart failure (New York Classification III-IV) or unstable angina pectoris within the last 6 months, or psychiatric illness that would limit compliance with study requirements as well as any condition that would preclude a participant from undergoing leukapheresis (e.g., within the previous 6 months: myocardial infarction, interventional cardiology procedure such as angioplasty or stent placement, pulmonary embolism or deep vein thrombosis).
* 13. Hypogonadal (T <175 ng/dL) or on continuous testosterone replacement therapy
* 14. Positive serology for HIV-1, HIV-2 or human T-lymphotropic virus (HTLV)-1, HTLV-2
* 15. Active hepatitis B or C
* 16. Any medical intervention, any other condition, or any other circumstance which, in the opinion of the investigator or the sponsor's Medical Monitor, could compromise adherence with study requirements or otherwise compromise the study's objectives.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males with proven adenocarcinoma of the prostate
Enrollment: 532 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadeem Sheikh, PhD, Study Director — Dendreon Pharmaceuticals, LLC
Locations (56):
- United States (56):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Arizona Institute of Urology, Tucson, Arizona
  - Urological Associates of Southern Arizona - East Office, Tucson, Arizona
  - Arkansas Urological Associates, PA, Little Rock, Arkansas
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - University of California Irvine, Orange, California
  - John Wayne Cancer Institute, Santa Monica, California
  - Skyline Urology, Torrance, California
  - University of Colorado Hospital Anschutz Cancer Pavilion, Aurora, Colorado
  - The Urology Center of Colorado, Denver, Colorado
  - Foothills Urology- Golden Office, Golden, Colorado
  - Advanced Urology Institute, Daytona Beach, Florida
  - Advanced Urology Institute of Georgia, Roswell, Georgia
  - Cook County Health, Chicago, Illinois
  - Rush University, Chicago, Illinois
  - Research by Design, Chicago, Illinois
  - Gottlieb Memorial Hospital, Glenview, Illinois
  - NorthShore University HealthSystem, Glenview, Illinois
  - Advanced Urology Associates, Joliet, Illinois
  - Comprehensive Urologic Care, Lake Barrington, Illinois
  - First Urology, Jeffersonville, Indiana
  - Iowa Clinical Research Corp., West Des Moines, Iowa
  - Kansas City Urology Care, PA, Overland Park, Kansas
  - Wichita Urology Group Research, Wichita, Kansas
  - Tulane University, New Orleans, Louisiana
  - Regional Urology, LLC, Shreveport, Louisiana
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Chesapeake Urology, Towson, Maryland
  - A. Alfred Taubman Health Care Center, Ann Arbor, Michigan
  - Michigan Institute of Urology, PC, Troy, Michigan
  - The Urology Group, Southaven, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Adult Pediatric Urology and Urogynecology - Omaha, Omaha, Nebraska
  - Urology Cancer Center and GU Research Network, Omaha, Nebraska
  - Delaware Valley Urology, Mount Laurel, New Jersey
  - Integrated Medical Professionals, PLLC, Melville, New York
  - Mount Sinai Health System, New York, New York
  - Associated Medical Professionals of NY, PLLC (AMP), Syracuse, New York
  - Associated Urologists of North Carolina - Raleigh, Raleigh, North Carolina
  - The Urology Group - Norwood Campus, Cincinnati, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Urology Institute Research, Springfield, Oregon
  - Urologic Consultants of Southeastern Pennsylvania, Bala-Cynwyd, Pennsylvania
  - Lancaster Urology, Lancaster, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - The Conrad Pearson Clinic, Germantown, Tennessee
  - Urology Associates, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - Urology San Antonio, San Antonio, Texas
  - Virginia Urology, Richmond, Virginia
  - Urology of Virginia, Virginia Beach, Virginia
  - Virginia Mason Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: Sipuleucel-T: Sipuleucel-T is an autologous cellular immunotherapy available as a suspension for intravenous infusion. Subjects randomized to sipuleucel-T arm will receive 3 infusions of sipuleucel-T at approximately 2-week intervals.
  sipuleucel-T: Sipuleucel-T is an autologous cell product consisting of antigen presenting cells (APCs) loaded with PA2024, a recombinant fusion protein composed of prostatic acid phosphatase (PAP), linked to granulocyte-macrophage colony-stimulating factor (GM-CSF).
- Control Arm: Active Surveillance: Subjects randomized to the control arm will be followed on Active Surveillance described in the schedule of events.
Period: Overall Study
Arm/Group | Treatment Group: Sipuleucel-T | Control Arm: Active Surveillance
Started | 356 | 176
Completed | 262 | 118
Not Completed | 94 | 58
Not completed — Withdrawal by Subject | 52 | 32
Not completed — Lost to Follow-up | 23 | 19
Not completed — Adverse Event | 1 | 0
Not completed — Death | 10 | 5
Not completed — Progressive Disease | 1 | 1
Not completed — Noncompliance | 1 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Screen fail post-randomization | 1 | 0
Not completed — Protocol Violation | 3 | 0
Not completed — No data available | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group: Sipuleucel-T | Control Arm: Active Surveillance | Total
Number analyzed (Participants) | 356 | 176 | 532
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 183 | 92 | 275
  >=65 years | 173 | 84 | 257
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (7.27) | 63.9 (7.72) | 64.0 (7.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 356 | 176 | 532
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 0 | 4
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 38 | 21 | 59
  White | 309 | 152 | 461
  More than one race | NA — This data point was not collected | NA — This data point was not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 2 | 3 | 5
Height [Mean (Standard Deviation); unit: centimeters] — Population: 3 participants did not report a baseline value for Height
  centimeters
    number analyzed (Participants) | 353 | 176 | 529
    (all) | 177.4 (6.7) | 178.1 (7.7) | 177.6 (7.1)
Weight [Mean (Standard Deviation); unit: kilograms] — Population: 3 participants did not report a baseline value for Weight
  kilograms
    number analyzed (Participants) | 353 | 176 | 529
    (all) | 91.6 (16.7) | 91.7 (20.0) | 91.7 (17.9)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: 3 participants did not report a baseline value for Weight in order to calculate the BMI
  kg/m^2
    number analyzed (Participants) | 353 | 176 | 529
    (all) | 29.1 (5.0) | 28.8 (5.4) | 29.0 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Sipuleucel-T Measured as the Percentage of Subjects Without Histological Reclassification (Gleason Group Upgrade).
Description: Percentage of participants without histological reclassification (Gleason group upgrade) within 36 months of randomization as determined by Blinded Independent Central Review (BICR)
  o Upgrade is defined as participants at randomization with either International Society of Urological Pathology (ISUP) Grade Group 1 (Gleason 3+3) upgraded to Grade Group 2 (Gleason 3+4) or higher or participants at randomization with Grade Group 2 upgraded to Grade Group 3 (Gleason 4+3) or higher.
Time Frame: Once all participants have completed at least 3 years following randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group: Sipuleucel-T | Control Arm: Active Surveillance
Number analyzed (Participants) | 356 | 176
Participants | 108 | 48
Statistical Analysis 1: Comparison: Treatment Group: Sipuleucel-T; Test type: Superiority; p = 0.4586, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.78 to 1.74]

ADVERSE EVENTS:
Time Frame: 4 years, 5 months
Description: All participants who received at least 1 infusion of sipuleucel-T (N=345) or after randomization in the control arm (N=176) were followed for safety.
  Total no. affected (74 in sipuleucel-T arm and 22 in Control arm) = the number of participants who experienced at least one serious adverse event (SAE). Participants may have had > 1 SAE. Total no. of SAEs may exceed the no. affected. Participants with <1 occurrence of the same event are counted only once.
Arm/Group | Treatment Group: Sipuleucel-T | Control Arm: Active Surveillance
All-Cause Mortality (participants affected / at risk) | 10/356 | 5/176
Serious Adverse Events (participants affected / at risk) | 74/345 | 22/176
Other Adverse Events (participants affected / at risk) | 321/345 | 133/176
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group: Sipuleucel-T (N=345) | Control Arm: Active Surveillance (N=176)
Haematuria (Renal and urinary disorders) | 4 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Coronary artery disease (Cardiac disorders) | 3 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Sepsis (Infections and infestations) | 3 | 1
Cellulitis (Infections and infestations) | 3 | 0
Peritonsillar abscess (Infections and infestations) | 2 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Syncope (Nervous system disorders) | 0 | 1
Aortic dissection (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina unstable (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Coronary ostial stenosis (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
COVID-19 (Infections and infestations) | 0 | 1
Cat scratch disease (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Pelvic infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
B-cell small lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dedifferentiated liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diffuse large B-cell lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Liposarcoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Paraganglion neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Peptic ulcer perforation (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 | 0
Death (General disorders) | 5 | 1
Adverse drug reaction (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1
Diabetic coma (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Myasthenia gravis (Nervous system disorders) | 1 | 0
Myelopathy (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Vertebrobasilar artery dissection (Nervous system disorders) | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Bipolar I disorder (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Hypoaesthesia (Skin and subcutaneous tissue disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Troponin increased (Investigations) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group: Sipuleucel-T (N=345) | Control Arm: Active Surveillance (N=176)
Chills (General disorders) | 70 | 2
Fatigue (General disorders) | 61 | 6
Erectile dysfunction (Reproductive system and breast disorders) | 39 | 19
Headache (Nervous system disorders) | 38 | 3
Paraesthesia (Nervous system disorders) | 38 | 0
Pyrexia (General disorders) | 38 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 34 | 8
Nausea (Gastrointestinal disorders) | 30 | 4
COVID-19 (Infections and infestations) | 29 | 9
Influenza like illness (General disorders) | 25 | 2
Haematuria (Renal and urinary disorders) | 22 | 10
Paraesthesia oral (Nervous system disorders) | 21 | 0
Diarrhoea (Gastrointestinal disorders) | 20 | 7
Dizziness (Nervous system disorders) | 20 | 6
Hypertension (Vascular disorders) | 20 | 9
Nocturia (Renal and urinary disorders) | 20 | 12
Pain (General disorders) | 20 | 0
Pollakiuria (Renal and urinary disorders) | 20 | 9
Rectal examination abnormal (Gastrointestinal disorders) | 20 | 6
Nasopharyngitis (Infections and infestations) | 18 | 2
Urinary tract infection (Infections and infestations) | 13 | 10
Prostatitis (Reproductive system and breast disorders) | 6 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the Study may be published and/or presented in an integrated manner reflecting the results observed across all participating centers. Accordingly, decisions on timing and content of publications and presentations relating to the Study will be coordinated by Dendreon in communication with institutions contributing patients to the Study.

DOCUMENTS (2):
  • Study Protocol (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/83/NCT03686683/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-17): https://cdn.clinicaltrials.gov/large-docs/83/NCT03686683/SAP_001.pdf